CLINICAL TRIAL: NCT02659917
Title: Performance of Glass-ionomer Cements in the Pit and Fissure Sealing and Atraumatic Restorative Treatment: a Randomized 2-year Clinical Trial
Brief Title: Performance of Glass-ionomer Cements: 2-year Follow-up
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fernanda Miori Pascon (Other)
Responsible Party: Sponsor-Investigator, Fernanda Miori Pascon, Teacher, University of Campinas, Brazil
Organization: University of Campinas, Brazil (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 3
Record Dates: First submitted 2016-01-12; First posted 2016-01-21 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: Dental Caries
Keywords: glass-ionomer cement; atraumatic restorative treatment; pit and fissure sealants
MeSH Terms: conditions — Dental Caries; Van der Woude syndrome | interventions — glass ionomer; Glass Ionomer Cements

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Ketac Molar® (3M/ESPE) - Glass ionomer (Active Comparator): Pit and fissure sealing using conventional glass-ionomer cement
  Interventions: Other: Glass ionomer
- Maxxion® (FGM) - Glass ionomer cement (Experimental): Pit and fissure sealing using conventional glass-ionomer cement
  Interventions: Other: Glass ionomer cement
- Ketac Molar® (3M/ESPE) - Glass ionomer - (Active Comparator): Restoration using conventional glass-ionomer cement
  Interventions: Other: -Glass ionomer-
- Maxxion® (FGM) - Glass ionomer cement - (Experimental): Restoration using conventional glass-ionomer cement
  Interventions: Other: -Glass ionomer cement-

INTERVENTIONS:
Other: Glass ionomer — Application of preventive agent
  Arms: Ketac Molar® (3M/ESPE) - Glass ionomer
Other: Glass ionomer cement — Application of preventive agent
  Arms: Maxxion® (FGM) - Glass ionomer cement
Other: -Glass ionomer- — Atraumatic Restorative Treatment
  Arms: Ketac Molar® (3M/ESPE) - Glass ionomer -
Other: -Glass ionomer cement- — Atraumatic Restorative Treatment
  Arms: Maxxion® (FGM) - Glass ionomer cement -

SUMMARY:
The purpose of this randomized clinical trial was evaluate the performance of two conventional glass-ionomer cements in the pit and fissure sealing and atraumatic restorative treatment in high caries risk children.

DETAILED DESCRIPTION:
Sealants were applied on sound permanent first molars by "press finger technique" and carious deciduous molars that required either class I or class II restorations were restored according to manufacturers' recommendations in order to caries prevention and control.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers that having at least two permanent first molars of opposite sides of the mouth, erupted in the oral cavity, caries-free and high-risk disease (presence of white spots, history of caries, plaque in smooth surfaces and gingivitis);
* Children who had one or two bilateral matched pairs of carious deciduous molars that required either class I or class II restorations.

Exclusion Criteria:

* Children who did not meet the minimum requirements for the achievement of sealants or parents / guardians did not agree to participate;
* No history of spontaneous pulpal pain.

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 147 (Actual)
Dates: Start 2008-08; Primary Completion 2009-02 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Number of the teeth with glass-ionomer cement retention and prevention of caries. | 6-month
  Criteria established by Frencken et al. (1998) was used.
Number of the teeth with good restoration and caries absence. | 6-month
  Criteria established by Frencken et al. (1998) was used.

SECONDARY OUTCOMES:
Frequency of loss of the sealing material and prevention of caries. | 6-month
  Criteria established by Frencken et al. (1998) was used.

CONTACTS AND LOCATIONS:
Overall Officials: Raquel V Rodrigues, PhD Student, Principal Investigator — Piracicaba Dental School - University of Campinas; Ana Carolina G Luciano, DDS, Principal Investigator — Piracicaba Dental School - University of Campinas; Kelly MS Moreira, MS Student, Principal Investigator — Piracicaba Dental School - University of Campinas

IPD SHARING:
Plan to Share IPD: No